CLINICAL TRIAL: NCT00200720
Title: Metabolic Consequences of High and Low Carbohydrate Diets
Brief Title: Effectiveness of a Low Carbohydrate Diet Versus a High Carbohydrate Diet in Promoting Weight Loss and Improved Health
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT000525-01 (NIH); R21AT000525-01 (NIH); 1R01AT001930 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2008-02

CONDITIONS: Obesity; Hypertension
Keywords: Diet; Carbohydrates; Weight Loss
MeSH Terms: conditions — Obesity; Hypertension; Weight Loss | interventions — Diet, High-Protein Low-Carbohydrate; Diet, Carbohydrate-Restricted; Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atkins Diet (Experimental): Participants randomized to this arm will consume a low carbohydrate diet as described by Dr. Robert Atkins in his book: Dr. Atkins' New Diet Revolution New York: Avon Books, 2002.
  Interventions: Behavioral: Atkins diet (low carbohydrate diet)
- DASH Diet (Active Comparator): Participants randomized to this arm will consume the Dietary Approaches to Stop Hypertension (DASH) diet as described here: http://www.nhlbi.nih.gov/health/public/heart/hbp/dash/new_dash.pdf
  Interventions: Behavioral: DASH diet (high carbohydrate diet)

INTERVENTIONS:
Behavioral: Atkins diet (low carbohydrate diet)
  Arms: Atkins Diet
Behavioral: DASH diet (high carbohydrate diet)
  Arms: DASH Diet

SUMMARY:
This study will examine the effects of a low carbohydrate diet versus a high carbohydrate diet on weight loss.

DETAILED DESCRIPTION:
The number of overweight and obese Americans has increased significantly in recent years. There are now many different diet plans being promoted by doctors and the media. The Atkins diet, a low carbohydrate nutritional plan, is especially popular; its advocates claim that following the diet will result in long-term weight loss with no negative effects. Another diet, called the Dietary Approaches to Stop Hypertension (DASH) diet, is a high carbohydrate diet designed to help treat and prevent high blood pressure. However, more thorough investigation of these claims is needed. This study will compare the short- and long-term effects of the Atkins diet to the (DASH) diet. This trial will enroll overweight and obese participants.

This study will last 30 months and will comprise two phases. Participants will be randomly assigned to either the Atkins or DASH diet for 30 months. During Phase 1, all participants will undergo 6 months of weekly group therapy to encourage weight loss. Phase 2 is a weight loss maintenance phase. During Phase 2, participants will have monthly meetings with a therapist for weight loss support. Study visits will occur at study entry and at Months 3 and 30. At each study visit, weight measurements, blood and urine collection, and x-rays will occur to determine participants' weight loss, cardiovascular health, kidney function, and bone density.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 27 to 50
* Fasting glucose less than 126 mg/dl
* Total fasting cholesterol less than 260 mg/dl
* Total fasting triglycerides less than 400 mg/dl
* Permission of primary care provider to participate in the study
* Normal liver and kidney function
* Willing to modify diet and other health behaviors
* Willing to use an acceptable method of contraception for the duration of the study

Exclusion Criteria:

* Any medical condition that may make weight loss medically inadvisable
* Weigh more than 400 lbs
* History of kidney failure
* Current use of more than 3 blood pressure medications
* Change in blood pressure medications within 3 months prior to study entry
* Diagnosis of cardiovascular disease within 6 months prior to study entry
* Cancer diagnosis within 2 years of study entry. Participants with basal cell skin cancer are not excluded.
* History of psychiatric hospitalization within 2 years prior to study entry
* Consumption of more than three alcoholic drinks a day
* Type I or II diabetes
* Current use of hypolipidemics, antipsychotics, hypoglycemics, glucocorticoids, or thyroid medication
* Plan to move during study
* Current participation in another clinical trial
* Pregnancy or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2005-04; Primary Completion 2009-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Weight loss | monthly
  Excess weight loss (greater than 5 pounds a week)would trigger patient assessment.

SECONDARY OUTCOMES:
Risk of cardiovascular disease | Every six months
  Elevated lipids or rising blood pressure during six month safety assessments would trigger additional participant evaluation
bone health | end of study
kidney function | every six months
neuroendocrine mechanisms of hunger and satiety | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Njeri Karanja, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States